CLINICAL TRIAL: NCT00156494
Title: "Attitudes About Smoking" A Telephone Survey of Parents of Young Urban Children
Brief Title: Attitudes About Smoking: A Telephone Survey
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Halcyon Hill Foundation (Other); Rochester City School District (Unknown); The Children's Institute (Other)
Responsible Party: Jill S. Halterman, MD, MPH, Halcyon Hill Foundation
Other Study IDs: 10182
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study involves telephone surveys of parents of young urban children with and without asthma to assess attitudes about smoking including personal smoking bans in their homes and cars, and beliefs about public policies regarding smoking.

ELIGIBILITY:
Inclusion Criteria:

* Child with asthma OR a matched child without asthma from the Rochester City School District

Exclusion Criteria:

* Non-english speaking family / parent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parents of children in the Rochester City School District
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States